CLINICAL TRIAL: NCT06540235
Title: VIBRANT-VM: Vestibular Investigation of Bone-conducted Resonant Analysis of Time-constants in Patients With Vestibular Migraines
Brief Title: The Effect of Bone-Conducted Stimulation on Rotary Chair Time Constants in Patients With Vestibular Migraines
Acronym: VIBRANT-VM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Otolith Labs (Industry)
Collaborators: Dizzy and Vertigo Institute of Los Angeles (Unknown); Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: OLith10904
Record Dates: First submitted 2024-07-31; First posted 2024-08-06 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Vestibular Migraine
Keywords: Vestibular Migraine; Central velocity storage; Vestibular condition; Migraine Associated Vertigo

STUDY DESIGN:
Who Masked: Participant
Masking Description: The device setting order is randomized to the participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- Off low high (Experimental): Device order will start with the device turned on but stimulation off, then the low setting and then the high setting
  Interventions: Device: Otolith Device Active
- Off high low (Experimental): Device order will start with the device turned on but stimulation off, then the high setting and then the low setting
  Interventions: Device: Otolith Device Active
- Off off off (Placebo Comparator): Device will always be turned on but stimulation off to measure test-retest variability.
  Interventions: Device: Otolith Device Inactive

INTERVENTIONS:
Device: Otolith Device Active — The device will be providing different levels of stimulation hypothesized to affect the vestibular system
  Arms: Off high low; Off low high
Device: Otolith Device Inactive — The device will be providing no stimulation to measure test-retest
  Arms: Off off off

SUMMARY:
The goal of this clinical trial is to learn if the Otolith Labs device can improve vestibular function of subjects with vestibular migraine.

The main questions it aims to answer are:

* When the Otolith Labs device is on, are objective measures of the vestibular system better than when the device is off?
* When the Otolith Labs device is on are subjective measures of the vestibular system better than when the device is off?
* Are the objective measures related to the subjective measures?

Researchers will change the order of the device settings to ensure the changes aren't due to the order they are tested.

Participants will:

* Wear the Otolith Labs device while in a rotary chair at different settings for different tests. All of the rotary chair testing will take less than an hour.
* Answer questions about how the rotary chair testing made them feel for each test.
* Answer questions about their every-day susceptibility to motion sickness and about their vestibular migraine symptoms.

DETAILED DESCRIPTION:
This study is designed to investigate the effects of The Otolith Labs bone conduction device (BCD) on the vestibular system. In the context of this trial, the BCD was designed and developed to reduce the effects of external stimulation of the vestibular system. The eventual intended use of the device is for people who have vestibular disorders (e.g. Vestibular Migraine, Meniere's Disease) who may benefit from a device that can provide a normalizing response to an abnormal vestibular neural signal.

To better understand the functioning principles of the BCD, the investigators want to conduct standard clinical testing using a rotary chair, specifically

1. Step velocity testing (SVT) with the chair rotating and vision denied
2. Optokinetic testing (OKT) with the chair stationary and visual field moving

Published studies have demonstrated that a reduction in the vestibulo-ocular reflex (VOR) time constants during optokinetic and velocity step testing is correlated with improved motion sickness symptoms. The investigators aim to determine if the BCD similarly reduces the VOR time constant. A reduction in time constant has been shown to be strongly correlated with a reduced time constant of integration in the central velocity storage (a long time constant very strongly correlates with motion sensitivity and with the severity of vestibular migraine episodes.

In this study, the BCD is set at one of three settings- turned off, low power level, high power level, -while the participant is undergoing testing at 60 °/s (patient's own motion for step velocity testing, or projected image for OKT). The same test methodology and equipment shall be used for all participants. In total, 6 rotational tests - one clockwise rotation and one counterclockwise rotation at each of the three power settings, and 6 static tests - with the visual field moving left then right at each of the three power settings, will be conducted and the order of the high/low power settings will be randomized to the second/third set of SVT and OKT. The device is adjusted to a new power level a few seconds before initiating each SVT and OKT.

Eye movements will be tracked during the SVT and OKT to evaluate decay in amplitudes and frequency of nystagmus over time (typically around 15 seconds). Comparison will be made between the three power conditions to evaluate the effect of bone conduction stimulation on the vestibular sense stimulated by rotation.

The participant will be prompted to report on the Fast Motion Scale (FMS) - a simple, validated 20 point verbally reported numerical rating scale - prior to and following each chair session to gauge the momentary level of motion sickness perception. The FMS will be reported a total of 12 times per participant (pre- & post-rotary tests).

Participants will complete the Motion Sickness Sensitivity Questionnaire Short Form (MSSQ-SF) to determine their history of sensitivity to provocative motion. Participants will also complete the Vestibular Migraine Patient Assessment Tool and Handicap Inventory (VM-PATHI) to assess the correlation of the potential change in time constants and VOR gain to the perceived severity of their vestibular migraine condition.

ELIGIBILITY:
Inclusion Criteria:

* Definite or probable vestibular migraine
* Residing in the United States

Exclusion Criteria:

* Head injury (e.g. skull fracture, concussion) within the last six months
* Neurodegenerative disorder
* Recent use of specified medications
* History of:

  * Vestibular neuritis / labyrinthitis
  * Vestibular schwannoma or acoustic neuroma
  * Radiographically unexplored unilateral or sudden sensorineural hearing loss
* History of surgery to the skull base or head,
* Surgery to the middle ear in the past 6 months,
* Surgery to the inner ear (e.g. labyrinthectomy) at any time.
* Eye surgery within the previous 3 months
* Significant reported history of ear disease, intravenous ototoxic medications

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-08-27 (Actual); Primary Completion 2025-08-27 (Actual); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Reduction of time constant | 60 minutes
  Time constant of slow-phase saccade attenuation in rotary chair

SECONDARY OUTCOMES:
Motion sickness symptom | 60 minutes
  Fast Motion Scale (FMS: min 0 to max 20, where "0" indicates no sickness at all and "20" indicates frank sickness)
Vestibular migraine handicap | 60 minutes
  Vestibular Migraine Patient Assessment Tool and Handicap Inventory (VM-PATHI: min 0 to max 100, where "0" indicates no handicap at all and "100" indicates complete handicap)
Motion sickness experience | 60 minutes
  Motion Sickness Susceptibility Questionnaire Short-form (MSSQ-Short: min 0 to max 54, where "0" indicates never sick and "54" indicates frequently sick)

CONTACTS AND LOCATIONS:
Overall Officials: Didier Depireux, PhD, Principal Investigator — Otolith Labs
Locations (2):
- United States (2):
  - Dizzy and Vertigo Institute of Los Angeles, Beverly Hills, California
  - Medical University of South Carolina, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers.